CLINICAL TRIAL: NCT05849883
Title: Bioequivalence Study of 20 mg Omeprazole Capsules in Indonesia Healthy Subject
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT Kalbe Farma Tbk (Industry)
Collaborators: PT Pharma Metric Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 551/STD/PML/2020
Record Dates: First submitted 2023-02-08; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Drug Use
Keywords: Omeprazole; Bioequivalence Study
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: Randomized, single blind, single dose, 2-treatment, 3-sequence, 3-period partial replicate design study with one week washout period in 36 healthy subjects under fasting condition.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omeprazole 20 mg capsules (Experimental): Subjects were given a single dose of 20 mg omeprazole of either formulation (test or reference) with 240 ml of water
  Interventions: Drug: Omeprazole 20 mg Capsules
- Losec® 20 mg capsules (Active Comparator): Subjects were given a single dose of 20 mg omeprazole of either formulation (test or reference) with 240 ml of water
  Interventions: Drug: Omeprazole 20 mg Capsules

INTERVENTIONS:
Drug: Omeprazole 20 mg Capsules — Omeprazole belongs to a class of antisecretory compounds, the substituted benzimidazoles, that suppress gastric acid secretion by specific inhibition of the H+/K+ ATPase enzyme system at the secretory surface of the gastric parietal cell. Because this enzyme system is regarded as the acid (proton) pump within the gastric mucosa, omeprazole has been characterized as a gastric acid-pump inhibitor, in that it blocks the final step of acid production
  Other Names: Losec® 20 mg capsules

SUMMARY:
The study was conducted to investigate whether 20 mg omeprazole capsules manufactured by PT. Dankos Farma for PT. Hexpharm Jaya is bioequivalent to its reference product, 20 mg Losec® capsules manufactured by AstraZeneca AB, Sweden, imported by PT. AstraZeneca Indonesia.

DETAILED DESCRIPTION:
Thirty six healthy subjects were given a single dose of 20 mg omeprazole capsules or 20 mg Losec® capsules with 240 mL of water. Then the blood samples for omeprazole were drawn and analyzed using LCMS/MS. All subjects sample plasma were analyzed for pharmacokinetic evaluation.

ELIGIBILITY:
The inclusion criteria were healthy male or female subjects who/with:

* had read the subject information and signed informed consent documents
* age range from 18 - 55 years
* body mass index between 18-25 kg/m2
* had a normal electrocardiogram
* had the blood pressure within normal range (systolic 90-120 mmHg and diastolic 60-80 mmHg)
* had the heart rate within normal range (60 - 100 bpm)
* had absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening.
* accepted to use protection (condom) before any intercourse with their spouse throughout the study

Excluded from the study were:

* those who were pregnant and/or nursing women (for women).
* those with history of contraindication or hypersensitivity to omeprazole, or other proton pump inhibitor drugs or other ingredients in the drugs or a history of serious allergic reaction to any drug, a significant allergic disease, or allergic reaction.
* those with a history or presence of medical condition which might significantly influence the pharmacokinetic of the study drug, e.g. chronic gastrointestinal disease, diarrhea, gastric surgery, renal insufficiency, hepatic dysfunction or cardiovascular disease.
* those with a history or presence of any coagulation disorder or clinically significant hematology abnormalities.
* those who were using any medication (prescription or non-prescription drug, food supplement, herbal medicine), particularly the medication known to affect the pharmacokinetic of the study drug, within one week prior to the drug administration day.
* those who had participated in any clinical study within 3 months prior to the study (<90 days).
* those who had donated or lost 300 ml (or more) of blood within 3 months prior to the study.
* those who smoked more than 10 cigarettes a day
* those who were reactive to SARS CoV-2 test.
* those with a history of travelling to another city within the last 14 days
* those with a history of direct contact with a COVID-19 positive person in the subject's neighborhood
* those with a history or present of sore throat, fever (with temperature more than 37°C) or dyspnea with in the last 14 days
* those who were positive to HIV, HBsAg, and HCV tests (to be kept confidential).
* those with a history of drug or alcohol abuse within 12 months prior to screening for this study.
* those who were unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow up visits, poor venous access.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Ratio of Cmax | before dosing and at 15, 30, 45, 60, 75, 90, 105 minutes, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, and 10 hours after drug administration
  The ratio between maximum concentration of test drug and reference drug after drug administration
Geometric Mean Ratio of AUCt | before dosing and at 15, 30, 45, 60, 75, 90, 105 minutes, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, and 10 hours after drug administration
  The ratio between area under curve from 0 to 10 hours of test drug and reference drug

SECONDARY OUTCOMES:
Pharmacokinetics Parameter of Cmax | before dosing and at 15, 30, 45, 60, 75, 90, 105 minutes, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, and 10 hours after drug administration
  Maximum plasma concentration (Cmax)
Pharmacokinetics Parameter of AUCt | before dosing and at 15, 30, 45, 60, 75, 90, 105 minutes, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, and 10 hours after drug administration
  Area Under Curve from 0 to 10 hours (AUCt)

CONTACTS AND LOCATIONS:
Overall Officials: Frans D Suyatna, Principal Investigator — PT Pharma Metric Labs; I Gusti Putu Bagus Diana Virgo, Study Director — PT Pharma Metric Labs
Locations (1):
- PT Pharma Metric Labs, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Kim YK, Yoon S, Yu KS, Kim BH, Yim SV. A bioequivalence study of two omeprazole formulations in healthy male volunteers. Int J Clin Pharmacol Ther. 2016 Nov;54(11):928-934. doi: 10.5414/CP202580. PMID 27615007
- [Background] Cederberg C, Andersson T, Skanberg I. Omeprazole: pharmacokinetics and metabolism in man. Scand J Gastroenterol Suppl. 1989;166:33-40; discussion 41-2. doi: 10.3109/00365528909091241. PMID 2690330
- [Background] Oosterhuis B, Jonkman JH. Omeprazole: pharmacology, pharmacokinetics and interactions. Digestion. 1989;44 Suppl 1:9-17. doi: 10.1159/000200098. PMID 2691315
- [Background] Dubcenco E, Beers-Block PM, Kim LP, Schotland P, Levine JG, McCloskey CA, Bashaw ED. A Proton Pump Inhibitor in the Reformulation Setting: Bioequivalence and Potential Implications for Long-Term Safety. Clin Transl Sci. 2017 Sep;10(5):387-394. doi: 10.1111/cts.12475. Epub 2017 Jun 15. PMID 28618191
- See also: Related Info — https://asean.org/wp-content/uploads/2012/10/BE_Guideline_FinalMarch2015_endorsed_22PPWG.pdf
- See also: Related Info — https://database.ich.org/sites/default/files/E6_R2_Addendum.pdf
- See also: Related Info — https://www.accessdata.fda.gov/drugsatfda_docs/label/2012/019810s096lbl.pdf